CLINICAL TRIAL: NCT03431194
Title: Midodrine is Effective in Management of Intradialytic Hypotension Among Critically-ill Patients With Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Collaborators: New Jeddah Clinic Hospital (Industry)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, Lecturer of Internal Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN-14716
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; midodrine; intensive care unit
MeSH Terms: conditions — Acute Kidney Injury | interventions — Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- midodrine group (Active Comparator): Patients will receive midodrine tablets
  Interventions: Drug: midodrine
- placebo group (Placebo Comparator): Patients receive sugary oral tablets therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: midodrine — oral midodrine tablets 5 mg
  Arms: midodrine group
Drug: Placebo
  Arms: placebo group

SUMMARY:
The aim of this randomized trial was to assess the efficacy of oral midodrine tablets for the management of intradialytic hypotension among critically ill patients with acute kidney injury.

DETAILED DESCRIPTION:
In This open -label study, patients in ICU with acute kidney injury are randomized to either midodrine tablets or placebo. the number of intradialytic episodes and both systolic and diastolic blood pressure between both groups are compared. Mortality and adverse effects are monitored and compared as well.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients
* acute kidney injury
* age above 18 years
* documented hypotension during dialysis

Exclusion Criteria:

* packed red blood cells transfusion
* intravenous inotropes
* alteration of blood pressure medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-02-19 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Number of hypotensive episodes | 30 days from start of hemodialysis
  Number of hypotensive episodes

SECONDARY OUTCOMES:
mean systolic blood pressure | 30 days from start of hemodialysis
  compare mean systolic blood pressure between the two arms
mean diastolic blood pressure | 30 days from start of hemodialysis
  compare mean diastolic blood pressure between the two arms
Mortality in each arm | 30 days from start of hemodialysis
  Number of dead patients in each arm

IPD SHARING:
Plan to Share IPD: No